CLINICAL TRIAL: NCT06858436
Title: The Role of SGLT2 Inhibitors in Stroke-reperfusion Injury:A Multi-Center, Randomized, Open-Label, Controlled Trial
Brief Title: SGLT2 Inhibitor Utilization Re-perfusion Therapy
Acronym: SUPER
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Principal Investigator, Po-Lin Chen, Director, Taichung Veterans General Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCVGH-1134501F
Record Dates: First submitted 2025-02-07; First posted 2025-03-05 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Acute Ischemic Stroke From Large Vessel Occlusion
Keywords: reperfusion therapy; SGLT2 inhibitor; malignant edema and transformation hemorrhage
MeSH Terms: conditions — Anthrax | interventions — Canagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- study group (Experimental): Patients who are enrolled will be randomly assigned to either the study group. Receiving Canagliflozin 100mg QD before undergoing mechanical thrombectomy. The prescribed duration of Canagliflozin 100mg QD will be 14 days.
  Interventions: Drug: Canagliflozin 100mg
- control group (No Intervention): Patients who are enrolled will be randomly assigned to either the control group.
  Not receiving Canagliflozin before undergoing mechanical thrombectomy.

INTERVENTIONS:
Drug: Canagliflozin 100mg — receiving Canagliflozin 100mg QD
  Other Names: Canagliflozin
  Arms: study group

SUMMARY:
Background:

Reperfusion therapies, including intravenous rt-PA and mechanical thrombectomy, significantly improve outcomes in acute ischemic stroke. However, these interventions also increase the risk of hemorrhagic transformation and malignant edema. Preclinical studies have demonstrated that Canagliflozin, an SGLT2 inhibitor, reduces astrocyte swelling and brain edema in a transient middle cerebral artery occlusion (tMCAo) model. While SGLT2 inhibitors have shown neuroprotective effects in the acute phase of ischemic stroke, their potential to mitigate hemorrhagic transformation and malignant edema following reperfusion therapy in humans remains unexamined.

Aims:

This study aims to evaluate the effect of SGLT2 inhibitors on hemorrhagic transformation and malignant edema in patients undergoing reperfusion therapy for acute ischemic stroke.

Methods:

This is a multi-center, randomized, open-label, controlled study enrolling ischemic stroke patients aged 18 years or older who meet predefined inclusion and exclusion criteria. Participants will be randomized to receive Canagliflozin 100 mg once daily for 14 days or no additional treatment before undergoing mechanical thrombectomy. Clinical data collection will include baseline demographics, medical and medication history, NIHSS scores at admission and 24 hours post-reperfusion, stroke subtype, modified Thrombolysis in Cerebral Infarction (TICI) scores, laboratory results, and modified Rankin Scale (mRS) scores at discharge and 3 months post-stroke.

The primary outcome is to assess the association between Canagliflozin use and the severity of hemorrhagic transformation and malignant edema. Hemorrhagic transformation will be classified using the Heidelberg criteria, and malignant edema will be defined as a midline shift of ≥5 mm. Brain imaging, including CT scans at 24 hours post-intervention and additional scans as clinically indicated, will be reviewed by blinded radiologists. Brain MRA will also be performed to assess infarct size and edema progression.

Importance:

This study aims to explore the potential for repurposing SGLT2 inhibitors as a therapeutic strategy in acute ischemic stroke. If Canagliflozin is shown to reduce hemorrhagic transformation and malignant edema, it could offer a novel adjunctive treatment to improve patient outcomes following reperfusion therapy.

DETAILED DESCRIPTION:
Clinical Study Protocol The Role of SGLT2 Inhibitors in Stroke-Reperfusion Injury: A Multi-Center, Randomized, Open-Label, Controlled Trial Version 6.0 | Date: 2024-12-10

1. Study Overview 1.1 Study Objectives Evaluate the efficacy of Canagliflozin 100 mg daily versus no treatment in reducing hemorrhagic transformation and malignant edema following reperfusion therapy in acute ischemic stroke.

1.2 Study Design

* Type: Multi-center, randomized, open-label, controlled trial
* Blinding: Open-label
* Randomization: Yes
* Design: Parallel-group
* Treatment Duration: 14 days
* Study Period: 3 years (2025-2027)
* Study Sites: Two medical centers in Taiwan
* Dose Adjustment: No 1.3 Endpoints

Primary Efficacy Endpoints:

1. Occurrence of malignant edema
2. mRS at 3 months post-stroke
3. Mortality at 3 months

Secondary Efficacy Endpoints:

1. Hemorrhagic transformation
2. Parenchymal hematoma type 2
3. NIHSS at 24 hours
4. mRS at discharge
5. EQ-5D at 3 months
6. Infarct size on MRI
7. MMP-9 upregulation after EVT

Primary Safety Endpoint:

* Incidence of adverse events (AEs)

  2. Study Population 2.1 Inclusion Criteria
* Age ≥18 years
* Acute ischemic stroke with large vessel occlusion, confirmed by CT perfusion
* Scheduled for mechanical thrombectomy 2.2 Exclusion Criteria
* CKD stage 4/5 (eGFR <30 mL/min/1.73m² or dialysis)
* Current or recent (≤3 months) SGLT2i use
* Hypersensitivity to Canagliflozin
* Type 1 diabetes
* Pregnancy or lactation 2.3 Withdrawal Criteria
* Voluntary withdrawal at any time
* Investigator-initiated withdrawal due to safety concerns or non-compliance

  3. Study Procedures
* Enrollment: ~105 patients/year (total 315 participants)
* Randomization: Canagliflozin 100 mg QD vs. control (no treatment) before thrombectomy
* Assessments:

  o Pre- & Post-EVT: Arterial blood sampling
  * 24h Post-EVT: Brain dual-energy CT, NIHSS
  * Day 3-Discharge: Brain MRA
  * At Discharge: mRS assessment
  * 3 Months Post-Stroke: mRS, EQ-5D 3.1 Imaging & Biomarker Analysis
* Malignant Edema: Midline shift ≥5 mm or symptomatic swelling requiring decompressive craniectomy
* Hemorrhagic Transformation: Classified by Heidelberg criteria, assessed via CT at 24 hours
* Infarct Volume: Measured via MRI using the ABC/2 method
* MMP-9 Analysis: Blood collected pre-/post-EVT, analyzed via ELISA

  4. Safety & Adverse Event Reporting
* Physicians will oversee patient safety and medication management.
* Participants will have direct access to study personnel for AE reporting.
* AEs will be reported to the IRB per regulatory guidelines. 4.1 Adverse Events (AE) and Management

  1. Hypoglycemia (~4%)

     * Symptoms: Sweating, confusion, dizziness
     * Management: Monitor blood glucose levels and adjust diabetes medications as needed
  2. Genital Infections (10-11% in women, 4% in men) o Symptoms: Itching, pain, discharge

     o Management: Maintain proper hygiene and use antifungal treatments if necessary
  3. Urinary Tract Infections (UTIs) (~5%)

     o Symptoms: Painful urination, urgency, fever

     o Management: Increase fluid intake and use antibiotics if symptoms persist
  4. Dehydration (1-2%)

     o Symptoms: Thirst, dark-colored urine, dizziness

     o Management: Stay hydrated and avoid excessive intake of diuretics such as caffeine and alcohol
  5. Hypotension (1-2%) o Symptoms: Dizziness, fainting, fatigue o Management: Monitor blood pressure, stay hydrated, and avoid sudden posture changes

  5. Criteria for Trial Termination

The trial may be stopped if:

* Safety concerns: Unexpected SAEs or high AE incidence outweighs benefits
* Regulatory issues: Recommendations from IRB/DSMB
* Operational issues: Insufficient enrollment or funding
* Interim analysis: Evidence of harm or lack of benefit

  6. Statistical Considerations 6.1 Sample Size
* Total required: 314 participants (157 per group)
* Power: 80%
* Alpha: 0.1 (one-sided) 6.2 Statistical Analysis
* Categorical Data: Fisher's exact test or χ² test
* Continuous Data: Mann-Whitney U-test, independent t-test
* Kaplan-Meier plots: Cumulative risk analysis
* Cox Proportional-Hazards Model: Malignant edema & hemorrhagic transformation incidence
* Repeated Measures ANOVA: NIHSS score changes
* Significance:

  o p < 0.1 (*); p < 0.05 (**) 6.3 Population for Analysis
* Intent-to-treat (ITT) for efficacy & safety assessments 6.4 Data Handling
* Poor-quality/missing data will be excluded.
* Protocol deviations will be documented and justified.

  7. Ethical & Regulatory Considerations 7.1 Ethical Approval & Patient Rights
* IRB Approval: Required before initiation
* Informed Consent: Participants will receive detailed study information and can withdraw at any time
* Data Security: Encrypted storage at two hospitals, access restricted to investigators 7.2 Data Access
* IRB permitted access for monitoring, audits, and inspections

  8. Funding & Insurance
* Funding: Provided by Veterans General Hospital
* Insurance: Coverage provided for participants due to study interventions

  9. References Key literature supporting Canagliflozin's neuroprotective potential in ischemic stroke and reperfusion injury.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have been diagnosed with acute ischemic stroke and large vessel occlusion by a neurologist, with confirmation supported by CT perfusion scans.
* Patients must be scheduled to undergo mechanical thrombectomy.

Exclusion Criteria:

* Patients with have stage 4 or 5 chronic kidney disease (estimated glomerular filtration rate (eGFR) below 30 mL/min/1.73 m² on dialysis)
* Patients with currently taking an SGLT2i or within 3 months prior to enrollment
* Patients with a known hypersensitivity or allergic reaction to Canagliflozin
* Patients with type 1 diabetes mellitus
* Patients with pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-01-23 (Estimated); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of malignant edema | On the 3rd to 5th day for MRI after EVT
  Diagnosed if midline shift ≥5 mm on brain imaging or symptomatic brain swelling requiring decompressive craniectomy, leading to in-hospital death, or coma at discharge.
mRS at 3rd month after stroke onset | 3 months after stroke onset
  Assesses health-related quality of life using modified Rankin Scale (mRS) to assess disability level post-stroke for understanding the recovery situation of the patient.
Mortality rate at 3rd month after stroke onset | After stroke onset in 3 months.
  To understand if the patient is surviving or not after stroke onset.

SECONDARY OUTCOMES:
Occurrence of hemorrhagic transformation | During hospitalization for 14 days
  Classified using the Heidelberg criteria to categorize hemorrhagic changes post-EVT.
Occurrence f parenchymal hematoma type2 | During hospitalization for 14 days
  Identified based on brain imaging and classified using the Heidelberg criteria, indicating severe hemorrhagic transformation.
NIHSS 24 hours later | 24 hours after EVT
  Neurological status assessed using National Institutes of Health Stroke Scale (NIHSS) to measure stroke severity and potential deterioration by neurologist.
mRS at discharge | Day 14 at hospital discharge
  Functional outcome evaluated using modified Rankin Scale (mRS) to assess disability level post-stroke.
EQ-5D at 3rd month after stroke onset | 3 months after stroke onset
  EQ-5D will be assessed three months after the onset of stroke through either face-to-face interviews or virtual platforms. Assesses health-related quality of life for understanding the recovery situation of the patient.
infarct size on brain MRI | Day 1 after EVT
  Measured using diffusion-weighted imaging (DWI), defined as a hyperintense area on b = 1000 mm/s² images.
  Calculation Method: ABC/2 method for infarct volume quantification.
upregulation of arterial biomarkers (MMP-9) after EVT | Day 1 before EVT is executed and after EVT finished
  Arterial blood will be collected from the puncture site, in a BD Vacutainer® EDTA tube, before and after EVT and centrifuged at 1,500 × g for 15 min at 4°C. The supernatant was collected as blood plasma. The level of MMP-9 in the plasma was measured following the manufacturer's protocol for the human MMP-9 Quantikine ELISA kit.

OTHER OUTCOMES:
Occurrence of adverse events as assessed by CTCAE v5.0 | During hospitalization for 14 days
  To understand if the patient have any occurrence of AE or SAE during the session.
  The result of finding any of the diseases listed on the CTCAE v5.0 will be reported to IRB of Taichung Veterans General Hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Po-Lin Chen, Study Director — Taichung Veterans General Hospital